CLINICAL TRIAL: NCT04523233
Title: Maternal Plasma/Urine/Hair/Amniotic Fluid Levels of Selected Trace Elements and Heavy Metals in Pregnancies Complicated With Neural Tube Defects
Brief Title: Metals/Vitamins Levels in NTD
Acronym: NTD&HMs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Collaborators: The Scientific Research Project Fund of Yozgat Bozok University (Unknown)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH8
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Neural Tube Defects
MeSH Terms: conditions — Neural Tube Defects | interventions — Amniocentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neural tube defects (NTDs): NTDs are a group of birth defects in which an opening in the spine or cranium remains from early in human development. Neural tube defects may be diagnosed during the ultrasound scan that is carried out around week 12 of the pregnancy or, more likely, during the anomaly scan that is carried out at around weeks 19 to 20.
  Interventions: Diagnostic Test: Amniocentesis
- Control group: The control group will be included pregnant women with healthy fetuses (n = 70), who were matched for gestational weeks and maternal age and underwent amniocentesis because of age-related risk or increased risk in the triple test.
  Interventions: Diagnostic Test: Amniocentesis

INTERVENTIONS:
Diagnostic Test: Amniocentesis — Amniocentesis is a procedure in which amniotic fluid is removed from the uterus for testing or treatment.
  Other Names: elements/vitamins concentrations measurements

SUMMARY:
Introduction: Heavy metals important pollutants produced from anthropogenic activities, has been suggested to be embryotoxic and fetotoxic in a lot of studies. The aims of this study were to determine the levels of trace elements and heavy metals, namely folic acid, zinc (Zn), molybdenum (Mo), vanadium (V), strontium (Sr), aluminium (Al), tin (Sn), antimony (Sb), mercury (Hg), calcium (Ca), iron ( Fe), magnesium (Mg), phosphorus (P), barium (B) and selenium (Se), in the amniotic fluid of pregnant women, and to investigate their relationship with neural tube defects (NTDs).

Methods: The study will be included 70 pregnant women whose fetuses were complicated with NTDs (study group) and 70 pregnant women with unaffected healthy fetuses (control group). The samples levels of elements and vitamins will be measured using inductively coupled plasma-mass spectrometry and will be compared between the two groups.

DETAILED DESCRIPTION:
Detailed Description:

This observational case-control study will be conducted at the Department of Obstetrics and Gynecology, Cengiz Gokcek Public Hospital, Gaziantep, Turkey, between August 2020 and March 2021. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (reference no: 2020/167). The study strictly will be adhered to the principles of the Declaration of Helsinki. All women will be provided written informed consent before the acquisition of all samples. The study will be included 140 pregnant women who underwent amniocentesis at the investigator's perinatology department.

The study group will be included 70 pregnant women whose fetuses were found to have congenital NTDs (eg, anencephaly, spina bifida, acrania, and encephalocele) on detailed ultrasonographic examinations between 16 and 37 weeks of pregnancy. The control group included pregnant women with healthy fetuses (n = 70), who were matched for gestational weeks and maternal age and underwent amniocentesis because of age-related risk or increased risk in the triple test. Then, this study will be determined maternal plasma/urine/hair, and amniotic fluid folic acid, zinc (Zn), molybdenum (Mo), vanadium (V), strontium (Sr), aluminium (Al), tin (Sn), antimony (Sb), mercury (Hg), calcium (Ca), iron ( Fe), magnesium (Mg), phosphorus (P), barium (B) and selenium (Se) concentrations in women with NTD compared to those of volunteer healthy pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women complicated with Neural tube defects
* Healthy pregnancy
* Singleton pregnancy

Exclusion Criteria:

1. pregnant women with any systemic condition (such as chronic hypertension, renal disease and )
2. women who have dyed their hair in the last 5 months
3. history of using any medication
4. presence of gestational hypertension or gestational diabetes
5. drug user
6. patients who had other fetal congenital abnormalities or genetic syndromes
7. multiple-gestation pregnancies
8. intrauterine fetal death
9. oligohydramnios

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: The study group included 70 pregnant women with congenital NTDs (e.g. anencephaly, spina bifida, acrania, NTDs, and encephalocele) with a normal karyotype, which were detected in detailed ultrasonographic examinations, and 70 healthy pregnancies will be selected for the control group.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
elements/vitamins concentrations in both group | 1 week
  The primary outcome in these analyses will compare folic acid, zinc (Zn), molybdenum (Mo), vanadium (V), strontium (Sr), aluminum (Al), tin (Sn), antimony (Sb), mercury (Hg), calcium (Ca), iron ( Fe), magnesium (Mg), phosphorus (P), barium (B) and selenium (Se) concentrations in NTD group and control group.

SECONDARY OUTCOMES:
compore in NTDs group | 1 week
  The secondary outcome in these analyses will compare the elements and vitamins concentrations in the spinal NTD group and the cranial NTD group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ovayolu A, Ovayolu G, Karaman E, Yuce T, Ozek MA, Turksoy VA. Amniotic fluid levels of selected trace elements and heavy metals in pregnancies complicated with neural tube defects. Congenit Anom (Kyoto). 2020 Sep;60(5):136-141. doi: 10.1111/cga.12363. Epub 2019 Nov 27. PMID 31743503
- [Result] Wilson RD; SOGC GENETICS COMMITTEE; SPECIAL CONTRIBUTOR. RETIRED: Prenatal screening, diagnosis, and pregnancy management of fetal neural tube defects. J Obstet Gynaecol Can. 2014 Oct;36(10):927-939. doi: 10.1016/S1701-2163(15)30444-8. PMID 25375307
- [Result] Yan L, Wang B, Li Z, Liu Y, Huo W, Wang J, Li Z, Ren A. Association of essential trace metals in maternal hair with the risk of neural tube defects in offspring. Birth Defects Res. 2017 Feb 15;109(3):234-243. doi: 10.1002/bdra.23594. PMID 27918138
- [Result] Nikolopoulou E, Galea GL, Rolo A, Greene ND, Copp AJ. Neural tube closure: cellular, molecular and biomechanical mechanisms. Development. 2017 Feb 15;144(4):552-566. doi: 10.1242/dev.145904. PMID 28196803

DOCUMENTS (1):
  • Study Protocol (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04523233/Prot_000.pdf